CLINICAL TRIAL: NCT02193568
Title: A Prospective, Single-Blinded, Randomized Study of Awake vs Intubated General Anesthesia in Patients Undergoing Elective Craniotomy for Supratentorial Glioma Resection
Brief Title: Light Sedation or Intubated General Anesthesia in Patients With Brain Cancer Undergoing Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, James Elder, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-12161; NCI-2014-01110 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-06-19; First posted 2014-07-17 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Adult Brain Tumor
Keywords: Supratentorial Glioma; Craniotomy
MeSH Terms: conditions — Brain Neoplasms | interventions — Anesthesia; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (light sedation) (Experimental): Patients receive light sedation (awake) and undergo craniotomy.
  Interventions: Procedure: Arm I (light sedation); Procedure: Arm II (intubated general anesthesia); Other: Arm II (intubated general anesthesia); Other: Arm I (light sedation)
- Arm II (intubated general anesthesia) (Active Comparator): Patients receive intubated general anesthesia and undergo craniotomy.
  Interventions: Procedure: Arm II (intubated general anesthesia); Other: Arm II (intubated general anesthesia); Procedure: Arm I (light sedation); Other: Arm I (light sedation)

INTERVENTIONS:
Procedure: Arm I (light sedation) — If patients experience excessive preoperative anxiety they will receive light sedation of midazolam 1 mg IV.In our standard practice, it is very rare that patients receive anxiolytic premedication for craniotomies, so it is unlikely that many will require midazolam. Two IVs will be placed, one for infusion of meds and one for possible resuscitation.
  Other Names: anesthesia
  Arms: Arm I (light sedation)
Procedure: Arm II (intubated general anesthesia) — Receive intubated general anesthesia
  Other Names: general anesthesia
  Arms: Arm II (intubated general anesthesia)
Procedure: Arm II (intubated general anesthesia) — Undergo craniotomy
  Other Names: therapeutic conventional surgery
Other: Arm II (intubated general anesthesia) — Ancillary studies
  Other Names: questionnaire administration
Procedure: Arm I (light sedation) — Undergo craniotomy
  Other Names: therapeutic conventional surgery
Other: Arm I (light sedation) — Ancillary studies
  Other Names: questionnaire administration

SUMMARY:
This randomized clinical trial studies light sedation compared with intubated general anesthesia (a loss of feeling and a complete loss of awareness that feels like a very deep sleep) in reducing complications and length of hospital stay in patients with brain cancer undergoing craniotomy. Craniotomy is an operation in which a piece of the skull is removed so doctors can remove a brain tumor or abnormal brain tissue. Light sedation allows patients to remain awake during their surgery, while intubated general anesthesia puts patients to sleep. Surgery complication rates may be reduced if intubated general anesthesia is avoided. Additionally, patients not receiving intubated general anesthesia tend to recover more quickly after surgery. It is not yet known whether light sedation is better at reducing complications and length of hospital stay compared to intubated general anesthesia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall hospital length of stay (LOS) in patients undergoing craniotomy with light sedation vs. general anesthesia.

SECONDARY OBJECTIVES:

I. To compare resource utilization between the two groups. II. To assess the frequency of post-operative delirium. III. To measure patient perceptions. IV. To track patient complications during hospital stay - nausea/vomiting, pain, hematology/lab stability, hemodynamic stability.

V. To track re-admission and extended hospital stay rates. VI. To compare cost of both approaches.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive light sedation (awake) and undergo craniotomy.

ARM II: Patients receive intubated general anesthesia and undergo craniotomy.

After completion of study, patients are followed up at 1month and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females
* Elective craniotomy for supratentorial brain tumors
* Primary brain cancer (presumed gliomas with no radiographic or clinical evidence of metastatic disease to the brain)
* First craniotomy
* American Society of Anesthesiologists (ASA) I-III
* Body mass index (BMI) < 35

Exclusion Criteria:

* Posterior fossa tumor/approach for tumor resection requiring the prone position
* Traumatic lesions/hematomas
* Emergency case
* Systemic disease burden with metastatic tumor to the brain
* Presence of medical co-morbidities, which, in the opinion of the investigator complicates the surgical procedure or would require additional hospital stay
* Necessity of awake procedure requiring intraoperative participation of patient due to the presence of the lesion in eloquent brain areas
* Prisoners
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04-30; Primary Completion 2016-10-08 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Compare overall hospital length of stay for patients in each of 2 arms | Up to 1 year
  Will be summarized for each arm and compared between light sedation and general anesthesia arm using two-sample test. Regression model will also be used to study the association between the length of stay and the type of anesthesia with potential confounder variables.

SECONDARY OUTCOMES:
Compare resource utilization between two groups | Up to 1 year
  Compare costs of hospital stay, anesthesia, and surgery
Assess the frequency of post-operative delirium | Up to 1 year
  Post-operative delirium will be assessed using the Memorial Delirium Assessment Scale (MDAS); a tool developed to measure the severity of delirium and reflects the main diagnostic criteria and symptoms of delirium. The MDAS is structured as a ten-item, four-point clinician-rated scale (possible range, 0-30) designed to quantify the severity of delirium in medically ill patients. A score of 13 has been recommended by the original authors as a cutoff for establishing the diagnosis of delirium.
Measure patient perceptions | Up to 1 year
  Will be measured by asking patients about their overall positive experiences, if they understood rationale behind non-intubated craniotomy; necessary to improve outcomes and minimize complications; self-protection/preservation, if they appreciated receiving information before surgery to help them make informed decisions, and their trust in the surgeon via survey to be conducted at the conclusion of the inpatient stay, before hospital discharge
Track patient complications during hospital stay | Up to 1 year
  Track patient nausea/vomiting, pain, hematology/lab stability, hemodynamic stability
Track re-admission and extended hospital stay rates | Up to 1 year from the date of surgery
  Tracking will be done using the EMR and follow-up calls

CONTACTS AND LOCATIONS:
Overall Officials: James Elder, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu